CLINICAL TRIAL: NCT01528332
Title: A Prospective, Randomized, Controlled, Double-Blind, Multi-Centre Study to Evaluate the Efficacy and Safety of Blue Light Therapy for Relief of Chronic Musculoskeletal Back Pain
Brief Title: Blue Light Device for Pain Therapy
Acronym: PAINCT02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philips Electronics Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAINCT02
Record Dates: First submitted 2012-02-01; First posted 2012-02-08 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Low Back Pain; Low Back Pain, Recurrent; Musculoskeletal Pain; Chronic Pain
Keywords: Musculoskeletal pain; Back pain; Chronic pain
MeSH Terms: conditions — Low Back Pain; Musculoskeletal Pain; Chronic Pain; Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pain Relief Patch (Experimental): Pain Relief Patch: Light wavelength 453 ± 7 nm, maximum 42 ± 6 mW/cm2 and average 20 ± 1 mW/cm², 30 minutes
  Interventions: Device: Pain Relief Patch
- Control PRP device (Active Comparator): Control PRP device: Light wavelength 531 ± 7 nm, maximum 0.4 ± 0.1 mW/cm² and average 0.2 ± 0.05 mW/cm², light on for 5 seconds, device worn for 30 minutes
  Interventions: Device: Control PRP device

INTERVENTIONS:
Device: Pain Relief Patch — The Pain Relief Patch is a non CE-marked device that is worn on the painful area of the back, where it shines light (453 ± 7 nm, maximum 42 ± 6 mW/cm2 and average 20 ± 1 mW/cm²). It will be used 5 times over 14 days for 30 minutes each time.
  Other Names: Blue light device, PRP patch, LED patch
  Arms: Pain Relief Patch
Device: Control PRP device — The Control PRP device is also a non CE-marked device. It is similar in appearance to the active Pain Relief Patch, except that it shines light of a different wavelength(531 ± 7 nm, maximum 0.4 ± 0.1 mW/cm² and average 0.2 ± 0.05 mW/cm²) for just 5 seconds before it turns off. Participants in the control arm will be treated with the control PRP device 5 times over 14 days for 30 minutes each time.
  Arms: Control PRP device

SUMMARY:
The purpose of this study is to determine if the Pain Relief Patch, which shines light of a limited wavelength on the painful area of the back, relieves chronic musculoskeletal back pain. At the same time, this study will gather information on side effects associated with use of the Pain Relief Patch. The study will compare the Pain Relief Patch to a patch that is similar in appearance, but which shines a different, presumed nontherapeutic, wavelength of light.

DETAILED DESCRIPTION:
This study will test the Pain Relief Patch (PRP), a new device containing LEDs that is to be worn on the skin of the painful area, to see if it is effective in relieving chronic musculoskeletal back pain. It will also test the safety of the patch. The LEDs in the PRP emit a certain kind of light (peak wavelength 453 nm) that stimulates the production of nitric oxide (NO) in the skin. NO has been shown to induce a number of actions that should contribute to pain relief, including relaxation of smooth muscle cells, dilation of blood vessels, increased concentrations of oxygen in the cells and washout of metabolic byproducts and toxins caused by cell injury or death. Participants in one treatment group will be treated 5 times over 2 weeks for 30 minutes with PRP patches in the clinic. Participants in the control arm will be treated for the same length of time with a similar device that contains LEDs that emit another wavelength of light that does not induce production of NO. To prevent the influence of expectations on the results, neither the participants nor the medical staff directly responsible for their treatment will be told with which of the test patches the participants are treated. Other clinic staff will be responsible for all activities that could identify treatment arm, including putting the devices on and removing them, and examining the condition of the participants' skin before and after treatment. To get an accurate measure of how effective the devices are, participants will score their pain several times before the treatment period begins, as well as before and after each treatment. They will also complete several pain questionnaires during the study.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 65 years of age, inclusive
* Is able to consent to participation by signing the informed consent form
* Has had localized mild to moderate (a score ≥ 2 and ≤ 6 on a 0 - 10 point pain intensity VAS) back pain for the 3 months prior to enrollment in study or longer
* Has a mean pain intensity VAS value (calculated from pain intensity VAS at Screening Visit, home assessment and pretreatment at Visit 1) between ≥ 2 and ≤6 at baseline prior to randomization
* Has skin type II, III or IV on the Fitzpatrick skin type scale (Types I - VI)
* Is willing and able to adhere to all study requirements, including accurate completion of VAS and questionnaires at the required time points, and is willing and able to travel to investigator's site to attend all required visits
* Is able to understand the study plan, its conditions, the therapy goals and expected outcomes

Exclusion Criteria:To be eligible for inclusion into this study, the patient must not meet any of the following criteria prior to enrollment:

General:

* Is participating in another clinical study at time of this study, or has participated in another study within the 30 days prior to signing the informed consent form
* Is pregnant or breast-feeding
* Is a sexually active female of childbearing potential and is not using a medically approved form of contraception
* Has moderate or severe arterial hypertension (WHO/ISH grade 2 or higher; systolic BP ≥ 160 and/or a diastolic BP ≥ 100), a history of stroke, myocardial infarction, angina pectoris, arteriosclerotic vascular disease (ASVD), or peripheral vascular disease, or (severe) congestive heart failure
* Is in poor general health
* Is an employee of the investigational site directly affiliated with this study and/or their immediate family members; an employee of the sponsor or the CRO

Back Pain Related:

* Has had any failed back surgery, or has had any surgery to torso, head or back within the previous 8 weeks
* Had an acute dislocation or fracture within the previous 8 weeks
* Has a degenerative central nervous system disease such as Multiple Sclerosis or Parkinson's disease; or a spinal stenosis that contributes to or is the cause of back pain; or Cauda equina syndrome, or other neurological symptoms indicating neuropathy
* Has any sensory deprivation or diagnosis of shingles or postherpetic neuralgia (specifically in mid-trunk region)
* Has wide spread pain
* Has any inflammatory disease that causes pain or any other chronic disease or infection known to cause pain (e.g. spondyloarthropathy, rheumatoid arthritis, Lupus erythematodes, Lyme borreliosis, etc.)
* Has schizophrenia, borderline syndrome or severe depression
* Has or has had cancer
* Has a history of severe osteoporosis (T score of 2.5 and a history of 1 or more bone fractures), or another severe bone disease
* Is unwilling to abstain from other non-drug back pain treatments, such as massage, sauna, transcutaneous electrical nerve stimulation, etc., for the duration of the trial
* Is unwilling to abstain from use of pain medication other than those recommended on steps 1 and 2 of the WHO Analgesic Ladder for the duration of the trial

Treatment Related:

* Has a known sun allergy, or known allergy to any device related material
* Uses steroids or any photosensitizing medication
* Has any known disease or idiopathic dermatosis such as porphyria, polymorphic light eruption, chronic actinic dermatitis, actinic prurigo or solar urticaria that causes photosensitivity
* Has a skin pathology, tattoo etc., or skin disease such as local infection, psoriasis, eczema etc. in the treatment area
* Has any anatomical pathology or other limitation that would prevent successful placement of the device
* Has an implanted medical device (screw, etc.) in or near the treatment area or an active implantable medical device such as cardiac pacemaker, defibrillator, neurostimulator, cochlear implant, active drug administration device anywhere in the body
* Is unwilling to abstain from sunbathing or use of tanning lights for the duration of the trial
* Is in the process of seeking early retirement, or is engaged in outstanding litigation involving back pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Bardenheuer, Prof. Dr., Principal Investigator — Clinic for Anaesthesiology and Supra-regional Centre of Pain Therapy and Palliative Care, University Hosp Heidelberg
Locations (3):
- Germany (3):
  - Clinic for Anaesthesiology and Supra-regional Center of Pain Therapy and Palliative Care, University Hosp Heidelberg, Heidelberg
  - Pain Therapy Section, Dept of Orthopedic Surgery and Traumatology, University Hosp Heidelberg, Heidelberg
  - University Medical Care Center Mannheim, Dept of Anaesthesiology and Surgical Care Medicine, Mannheim

REFERENCES:
- [Derived] Baron R, Morlion B, Dahan A, Uberall M, von Basum G, Wild I. A prospective, randomized, controlled, double-blind, multi-center study to evaluate the efficacy and safety of a blue light device for the treatment of chronic back pain. Front Pain Res (Lausanne). 2024 Jul 23;5:1444401. doi: 10.3389/fpain.2024.1444401. eCollection 2024. PMID 39109241

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of First Enrollment: 03-Feb-2012 Date of Last Patient Last Visit: 03-Jul-2012
Period: Overall Study
Arm/Group | Pain Relief Patch | Control PRP Device
Started | 85 | 86
Completed | 81 | 84
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Relief Patch | Control PRP Device | Total
Number analyzed (Participants) | 85 | 86 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 86 | 171
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (10.7) | 51.4 (8.3) | 50.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 30 | 28 | 58
Region of Enrollment [Number; unit: participants]
  Germany | 85 | 86 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Mean of Three Measurements at Screening, Prior to Treatment Visit 1 and Treatment Visit 1 Pretreatment) in the Average Visual Analog Scale (VAS) Pain Intensity Over the 5 Treatment Days
Description: Pain intensity scored on a 10.0 cm VAS with the endpoints 0 = no pain; 10 = worst pain imaginable
Time Frame: Baseline (Visit 1/day -7, at home and Visit 2/day +1), Treatment (Visits 2-6 post treatment/days +1 to +14)
Measure: Mean (Standard Error); unit: cm
Arm/Group | Pain Relief Patch | Control PRP Device
Number analyzed (Participants) | 85 | 86
cm | -1.24 (0.11) | -0.87 (0.11)

2. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) at Visit 5
Description: The RMDQ is a 24 list of yes/no questions about the effects of back pain on the participants daily activities. Each positive answer is a point; maximum total score = 24.
Time Frame: Baseline (days -7 to +1) to Treatment 5 (day +14)
Reporting Status: Not Posted

3. Secondary Outcome: Change From Baseline in VAS Pain Intensity at Follow up
Time Frame: Baseline (day -7 to 1) to Follow-up (up to day +42)
Reporting Status: Not Posted

4. Secondary Outcome: Change From Treatment in VAS Pain Intensity at Follow up
Time Frame: Treatment (day +1 to +14) to Follow-up (up to day +42)
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in RMDQ at Follow up
Time Frame: Baseline (days -7 to +1) to Follow-up (up to day +42)
Reporting Status: Not Posted

6. Secondary Outcome: Change From Treatment in RMDQ at Follow up
Time Frame: Treatment (days +1 to +14) to Follow up (up to day +42)
Reporting Status: Not Posted

7. Secondary Outcome: Frequency, Severity, Nature and Duration of Adverse Events During the Whole Duration of the Study
Description: Adverse events will be assessed using descriptive statistical methods and compared between treatment arms.
Time Frame: Baseline (days -7 to -1) to Follow up (up to day +42)
Reporting Status: Not Posted

8. Secondary Outcome: Vital Sign Parameters
Description: Vital signs (blood pressure and pulse)will be assessed at each visit and changes from baseline compared between the treatment groups
Time Frame: Baseline (days -7 to -1) to Follow up (up to day +42)
Reporting Status: Not Posted

9. Secondary Outcome: Changes From Baseline in Skin Condition
Description: Skin condition (erythema and hyperpigmentation as measured with the MX-18) and appearance (recorded with Polaroid photos) will be assessed once each at baseline and follow up, and before and after each treatment. The changes from baseline will be analysed using descriptive statistics and the two treatment arms compared.
Time Frame: Baseline (days -7 to -1) to Follow up (up to day +42)
Reporting Status: Not Posted

10. Secondary Outcome: Average Visual Analog Scale Pain Relief Over 5 Treatments
Description: The average pain relief scored on a 10.0 cm VAS pain relief scale (endpoints 0 = no pain, 10 = no relief
Time Frame: 5 treatments (days +1 to +14)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pain Relief Patch | Control PRP Device
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/86
Other Adverse Events (participants affected / at risk) | 62/85 | 60/86
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pain Relief Patch (N=85) | Control PRP Device (N=86)
Headache (Nervous system disorders) | 27 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
General Disorders (General disorders) | 17 | 12 — The frequency of the single terms is less than 5% for all terms within this group
Gastrointestinal disorders (Gastrointestinal disorders) | 11 | 15 — The frequency of the single terms is less than 5% for all terms within this group
Infections and Infestations (Infections and infestations) | 5 | 10 — The frequency of the single terms is less than 5% for all terms within this group
Ear and labyrinth disorders (Ear and labyrinth disorders) | 5 | 4 — The frequency of the single terms is less than 5% for all terms within this group
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 6 — The frequency of the single terms is less than 5% for all terms within this group
Psychiatric disorders (Psychiatric disorders) | 1 | 6 — The frequency of the single terms is less than 5% for all terms within this group
Back Pain (Musculoskeletal and connective tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No